CLINICAL TRIAL: NCT03838978
Title: Evaluation of the Calypso Knee System for Symptom Relief in Subjects With Medial Knee Osteoarthritis, OUS
Brief Title: Calypso Knee System Clinical Study, OUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moximed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP0002 (formerly CLIN102918)
Record Dates: First submitted 2019-02-11; First posted 2019-02-12 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Single Arm Study Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Calypso Knee System (Experimental): Calypso Knee System
  Interventions: Device: Calypso Knee System (Implantable Shock Absorber)

INTERVENTIONS:
Device: Calypso Knee System (Implantable Shock Absorber) — The Calypso Knee System is an extra-capsular knee implant designed to fill the therapeutic gap between conservative care and more invasive surgical interventions for knee osteoarthritis.
  Other Names: MISHA(R) Knee System

SUMMARY:
A study to evaluate the safety and effectiveness of the Calypso Knee System when used in subjects with symptomatic osteoarthritis of the medial compartment of the knee.

DETAILED DESCRIPTION:
Prospective, multicenter clinical study of the Calypso Knee System. A total of 81 subjects were enrolled in this study. Male or female subjects age 25 to 65 years, with a diagnosis of medial knee osteoarthritis and study knee pain with an overall WOMAC pain score ≥ 40 (scale 0-100).

The Calypso group was investigated under two clinical protocols, CP0001 in the USA, and CP0002 in Europe. Both clinical protocols followed the same supporting protocols and plans, such as radiographic, statistical, Clinical Events Committee (CEC), etc. The results from the combined analysis have been reported in both NCT03671213 (CP0001) and NCT03838978 (CP0002).

ELIGIBILITY:
Inclusion Criteria:

1. Participants age - 25 to 65 years
2. Body Mass Index (BMI) of < 35, Weight < 300 lbs (136 kg)
3. Knee osteoarthritis pain on the inner side of knee that has continued after at least 6 months of non-operative treatment

Exclusion Criteria:

1. Symptoms of osteoarthritis in the other knee or in lateral (outer) or patellofemoral compartments of the target knee
2. Knee ligament or meniscal instability
3. Other bone or joint conditions such as Rheumatoid arthritis, Paget's disease, Charcot's disease or general conditions such as allergy or hypersensitivity to certain metals, active infection, certain neurological conditions, use of medication such as steroids or chemotherapy that could impact study participation or results

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2025-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Flanigan, MD, Principal Investigator — Ohio State University
Locations (5):
- UZ Gent, Ghent, Belgium
- Poland (4):
  - SPORTO, Lodz
  - Zagiel Med Hospital, Lublin
  - Carolina Medical Center, Warsaw
  - Mirai Clinic, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Diduch DR, Crawford DC, Ranawat AS, Victor J, Flanigan DC. Implantable Shock Absorber Provides Superior Pain Relief and Functional Improvement Compared With High Tibial Osteotomy in Patients with Mild-to-Moderate Medial Knee Osteoarthritis: A 2-Year Report. Cartilage. 2023 Jun;14(2):152-163. doi: 10.1177/19476035231157335. Epub 2023 Feb 23. PMID 36823955

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Calypso Clinical Study enrolled 81 subjects in the investigational (Calypso) arm. The historical control arm (HTO) is from a prior Moximed sponsored clinical trial. The results presented include data from the historical control arm for comparison, per the protocol.
Groups:
- Calypso Knee System: Calypso Knee System: The Calypso Knee System is an extra-capsular knee implant designed to fill the therapeutic gap between conservative care and more invasive surgical interventions for knee osteoarthritis.
- High Tibial Osteotomy (HTO): Historical Control: HTO is a surgical treatment intended to reduce or eliminate pain and improve the function of a knee affected by medial compartment OA. All subjects underwent an open wedge osteotomy (OWO).
  The historical control arm (HTO) is from a prior Moximed sponsored clinical trial. The results presented include data from the historical control arm for comparison, per the protocol.
Period: Overall Study
Arm/Group | Calypso Knee System | High Tibial Osteotomy (HTO)
Started | 81 | 81
Completed | 73 | 65
Not Completed | 8 | 16

BASELINE CHARACTERISTICS:
Groups:
- High Tibial Osteotomy (HTO): Historical Control: HTO is a surgical treatment intended to reduce or eliminate pain and improve the function of a knee affected by medial compartment OA. All subjects underwent an open wedge osteotomy (OWO).
- Total: Total of all reporting groups
Arm/Group | Calypso Knee System | High Tibial Osteotomy (HTO) | Total
Number analyzed (Participants) | 81 | 81 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (7.71) | 52.5 (7.58) | 51.8 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 28 | 60
  Male | 49 | 53 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 78 | 50 | 128
  Unknown or Not Reported | 0 | 30 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 80 | 80 | 160
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (3.44) | 29.3 (4.36) | 28.8 (3.94)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite Clinical Success (CCS)
Description: A subject is considered a Composite Clinical Success (CCS), at 24 months, if the subject meets all of the following:
  1. Clinically significant improvement of at least 20% from baseline on the WOMAC pain questions in the KOOS Knee questionnaire with a change of ≥10 points
  2. Clinically significant improvement of at least 20% from baseline on the WOMAC function questions in the KOOS Knee questionnaire with a change of ≥10 points
  3. Freedom from the following device-related serious adverse events:
     * Deep infection requiring surgical intervention (Both arms)
     * Damage to adjacent neurovascular or ligament structures necessitating reconstruction (Both arms)
     * Non-union (HTO only)
  4. Maintenance of implant integrity as evaluated by radiographic assessment
  5. Endpoint Subsequent Surgical Intervention (SSI)
Time Frame: From baseline to 24 months
Measure: Number; unit: percentage of subjects
Groups:
- Calypso Knee System: The Calypso Knee System is an extra-capsular knee implant designed to fill the therapeutic gap between conservative care and more invasive surgical interventions for knee osteoarthritis.
Arm/Group | Calypso Knee System | High Tibial Osteotomy (HTO)
Number analyzed (Participants) | 81 | 81
percentage of subjects | 83.5 | 57.2
Statistical Analysis 1: Comparison: Calypso Knee System vs High Tibial Osteotomy (HTO); For missing data in both Arms/Groups, multiple imputation was performed for the primary CCS analysis; Test type: Superiority — Non-inferiority is demonstrated if the 90% LB > -10.0%. If non-inferiority was met, superiority could be tested. Superiority is demonstrated if 97.5% LB > 0.0%; Device group differences and two-sided 90% and 97.5% confidence interval lower bounds (LB) adjusting for propensity score (PS) subclass based on PS subclass weights (ATT). Noninferiority is demonstrated if the 90% LB > -10.0%. Superiority is demonstrated if 97.5% LB >0.0%. Two-sided 97.5% LB is evaluated rather than two-sided 95.0% LB since the superiority type 1 error is split between testing superiority in terms of Month 24 CCS and then separately for a set of superiority secondary endpoints with type 1 error control maintained through the use of Hochberg approach (following demonstration of non-inferiority)

2. Secondary Outcome: Time to Full Weight Bearing (Days)
Time Frame: Through study completion (number of days to full weight bearing)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Calypso Knee System | High Tibial Osteotomy (HTO)
Number analyzed (Participants) | 81 | 77
days | 13.4 (10.12) | 58 (39.91)

3. Secondary Outcome: WOMAC Pain Percent Change to Month 3
Description: The Knee Injury and Osteoarthritis Outcome Score (KOOS) Knee Survey includes the Western Ontario and McMasters University Osteoarthritis Index (WOMAC) in its complete and original format (with permission), and WOMAC scores can be calculated from the KOOS Knee questionnaire. The response to each question is summed and the resultant scores are transformed to a 0-100 scale. A WOMAC score of zero (0) represents no knee problems and one hundred (100) represents extreme knee problems.
Time Frame: From baseline to 3 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Calypso Knee System | High Tibial Osteotomy (HTO)
Number analyzed (Participants) | 81 | 72
percentage of change | -55.5 (29.3) | -33.4 (35.8)

4. Secondary Outcome: WOMAC Pain Percent Change to Month 24
Description: as for outcome 3
Time Frame: From baseline to 24 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Calypso Knee System | High Tibial Osteotomy (HTO)
Number analyzed (Participants) | 72 | 58
percentage of change | -76.0 (28.2) | -64.7 (33.0)

5. Secondary Outcome: WOMAC Function Percent Change to Month 3
Description: as for outcome 3
Time Frame: From baseline to 3 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Calypso Knee System | High Tibial Osteotomy (HTO)
Number analyzed (Participants) | 81 | 75
percentage of change | -52.2 (32.0) | -25.2 (37.0)

6. Secondary Outcome: WOMAC Function Percent Change to Month 24
Description: as for outcome 3
Time Frame: From baseline to 24 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Calypso Knee System | High Tibial Osteotomy (HTO)
Number analyzed (Participants) | 72 | 64
percentage of change | -73.9 (29.6) | -58.8 (35.8)

ADVERSE EVENTS:
Time Frame: Index procedure (enrollment) through 24 months (790 days)
Description: Serious Adverse Events reported as adjudicated as device and/or procedure related by the Clinical Events Committee (CEC).
Arm/Group | Calypso Knee System | High Tibial Osteotomy (HTO)
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/81
Serious Adverse Events (participants affected / at risk) | 18/81 | 39/81
Other Adverse Events (participants affected / at risk) | 20/81 | 14/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calypso Knee System (N=81) | High Tibial Osteotomy (HTO) (N=81)
Infection: Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infection: Deep (Infections and infestations) | 4 (4) | 2 (2)
Infection: Superficial incisional surgical site (Infections and infestations) | 0 (0) | 1 (1)
Anesthesia Complications: Other (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Discomfort: Catching or pulling sensations (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Discomfort: Inability to perform certain tasks (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hospital readmission: Removal of implant due to dissatisfaction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nerve injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Other: Other, bone consolidation (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain: Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 29 (30)
Scar formation: Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Scar formation: Periprosthetic adhesions/fibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Swelling: Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Wound: Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Wound: Wound dehiscence (post-explant) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Psychological event: Other (Psychiatric disorders) | 1 (1) | 0 (0)
Bleeding: Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis: Superficial Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calypso Knee System (N=81) | High Tibial Osteotomy (HTO) (N=81)
Nerve injury (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Pain: Pain (Musculoskeletal and connective tissue disorders) | 16 (18) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution agrees study is multi-center study conducted by Sponsor and agrees not to publish until study completion and not before publication of multicenter results in peer-reviewed journal. Thereafter, Institution may publish its site experience. Sponsor reserves exclusive right to publish results and establish authorship based on compliance, contribution and acceptance of responsibilities. If no publication submitted by Sponsor within 12 months of study closure, Institution may publish.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT03838978/Prot_SAP_000.pdf